CLINICAL TRIAL: NCT04727502
Title: Comparison of Duloxetine Versus Pregabalin in Post-mastectomy Pain Syndrome: a Randomized Controlled Trial
Brief Title: Comparison of Duloxetine Versus Pregabalin
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Cancer Institute, Egypt (Other)
Responsible Party: Principal Investigator, Mohammed Abdelfattah Abdelwadod, Mohammed Abdelfattah Abdelwadod, National Cancer Institute, Egypt
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AP2007-50104
Record Dates: First submitted 2020-12-25; First posted 2021-01-27 (Actual); Last update posted 2021-01-27 (Actual); Status verified 2021-01

CONDITIONS: Drug Effect
Keywords: pregabalin and Duloxetine
MeSH Terms: interventions — Duloxetine Hydrochloride

STUDY DESIGN:
Intervention Model Description: 2 equal groups ( Group A) :receive duloxetine for 12 weeks and (Group B) control group receive pregabalin for 12 weeks .
  • Dosing and administration Group A) Duloxetine 30 mg /day at bed time and (Group B) control group Pregablin 150mg /day( 75 mg /12 hours
Who Masked: Care Provider, Outcomes Assessor
Masking Description: Randomization is done using computer generated sequence. Concealment will be achieved by opaque envelope.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ( Group Duloxetine ) (Active Comparator): • Dosing and administration (Group A) Duloxetine 30 mg /day oral intake at bed time
  Interventions: Drug: Duloxetine
- (Group Pregablin ) (Active Comparator): control group Pregablin 150mg /day( 75 mg /12 hours ) oral intake.
  Interventions: Drug: Pregablin

INTERVENTIONS:
Drug: Duloxetine — duloxetine
  Arms: ( Group Duloxetine )
Drug: Pregablin — Pregablin
  Arms: (Group Pregablin )

SUMMARY:
Chronic post mastectomy pain syndrome (PMPS) is a chronic post-surgical neuropathic pain following breast cancer surgeries and lasting more than three months after surgeries. Pregabalin is originally used as an antiepileptic drug and identiﬁed as treatment for neuropathic pain .There are several recent reviews have revealed that it reduces post-operative opioid consumption and improves pain scores after breast surgeries. Duloxetine is a serotonin and norepinephrine reuptake inhibitor. Its mechanism of action is related to the potentiation of serotonergic and noradrenergic activity in the descending inhibitory pain pathways of the central nervous system and used for treatment of neuropathic pain conditions as painful diabetic neuropathy, neuropathic pain of lung cancer and chemotherapy induced sensory neuropathy

DETAILED DESCRIPTION:
Patients with of 3 months of chronic neuropathic pain after breast surgery (either modified radical mastectomy or conservative breast surgery) combined with axillary dissection is considered as post mastectomy pain syndrome which is defined as pain involving the anterior aspect of the chest, axilla, and/or upper arm with the classical features of neuropathic pain including numbness, tingling, burning, shooting, stinging, or stabbing pains, and hyperesthesia.

* They are divided to 2 equal groups: ( Group A) receive duloxetine for 12 weeks and (Group B) control group receive pregabalin for 12 weeks .
* Dosing and administration Group A) Duloxetine 30 mg /day at bed time and (Group B) control group Pregablin 150mg /day( 75 mg /12 hours )
* Randomization and blinding: Randomization is done using computer generated sequence. Concealment will be achieved by opaque envelope.
* Concomitant therapy :opioid therapy according to WHO step ladder in cancer pain

ELIGIBILITY:
Inclusion Criteria:

* Female, history of breast surgery and patients with post mastectomy pain

Exclusion Criteria:

* pregnancy,history of allergy to Pregabalin or duloxetine, pregnancy or lactation, history of pregabalin or gabapentin intake in the preceding three months, history of radiotherapy and history of drug abuse

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Adult female patients underwent breast cancer surgeries presented with post mastectomy pain syndrome
Enrollment: 70 (Estimated)
Dates: Start 2020-12-20 (Actual); Primary Completion 2021-03 (Estimated); Study Completion 2021-04 (Estimated)

PRIMARY OUTCOMES:
visual analogue score | baseline till 12 weeks of treatment
  visual analogue score with least pain score is 0 and worst pain is 10

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Abdel Wadod, MD, Principal Investigator — National Cancer Institute, Cairo University, Egypt
Locations (1):
- Nataional Cancer Instituite, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided